CLINICAL TRIAL: NCT02729597
Title: Tracking the Brain in Myotonic Dystrophies: a 5-year Longitudinal Follow-up Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: Forschungszentrum Juelich (Other); Life and Brain Center Bonn (Unknown); The Marigold Foundation (Unknown)
Responsible Party: Principal Investigator, Cornelia Kornblum, Prof. Dr., University Hospital, Bonn
Other Study IDs: DM-1-2
Record Dates: First submitted 2016-03-23; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Myotonic Dystrophy 1; Myotonic Dystrophy 2
Keywords: neuromuscular disorders; MRI; white matter; brain; myotonic dystrophy
MeSH Terms: conditions — Myotonic Dystrophy; Neuromuscular Diseases | interventions — Health Records, Personal; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Myotonic dystrophy type 1 patients: Patients with myotonic dystrophy type 1 (diagnosis confirmed by genetic testing) who meet all inclusion and exclusion criteria for patients.
  To be assessed at baseline and follow-up:
  medical history, neurological clinical examination, neuropsychological testing, brain MRI
  Interventions: Other: medical history; Other: neurological clinical examination; Other: neuropsychological testing; Other: brain MRI
- Myotonic dystrophy type 2 patients: Patients with myotonic dystrophy type 2 (diagnosis confirmed by genetic testing) who meet all inclusion and exclusion criteria for patients.
  To be assessed at baseline and follow-up:
  medical history, neurological clinical examination, neuropsychological testing, brain MRI
  Interventions: Other: medical history; Other: neurological clinical examination; Other: neuropsychological testing; Other: brain MRI
- Controls: Healthy control subjects who meet all inclusion and exclusion criteria for healthy controls.
  To be assessed at baseline and follow-up:
  medical history, neurological clinical examination, neuropsychological testing, brain MRI
  Interventions: Other: medical history; Other: neurological clinical examination; Other: neuropsychological testing; Other: brain MRI

INTERVENTIONS:
Other: medical history — The complete medical history (including cardiovascular risk factors and medication) will be assessed at baseline and follow-up.
Other: neurological clinical examination — Neurological examination will be performed at baseline and follow-up.
Other: neuropsychological testing — Neuropsychological testing using a 13 item test battery will be performed at baseline and follow-up.
Other: brain MRI — Brain MRI ( 3.0 T) will be performed using the same hard- and software at baseline and follow-up.

SUMMARY:
The natural history of brain affection in myotonic dystrophy types 1 and 2 is still unknown. The investigators designed a 5-year longitudinal neuropsychological and neuroimaging follow-up study to address this issue. Myotonic dystrophy type 1, myotonic dystrophy type 2 patients, and healthy controls were enrolled. All participants undergo clinical-neurological examinations, neuropsychological analyses according to a 13-item neuropsychological test battery, and 3T-brain MRI including voxel-based morphometry and diffusion tensor imaging at baseline and at follow-up using identical examination protocols.

DETAILED DESCRIPTION:
It is unknown whether brain affection in myotonic dystrophy types 1 and 2 is due to neurodevelopmental defects, neurodegeneration, or both. An exact definition of the nature and dynamic of brain affection is of urgent need for the identification of clinical trial outcome parameters and the design of therapy compounds. The investigators planned a 5-year longitudinal study to examine the natural history of functional and structural brain affection. Myotonic dystrophy type 1, myotonic dystrophy type 2 patients, and healthy controls were enrolled. All participants undergo clinical-neurological examinations, neuropsychological analyses according to a 13-item neuropsychological test battery, and 3T-brain MRI at baseline and at follow-up using identical examination protocols. The intended time span between baseline and follow-up examinations is 5 years minimum. To investigate gray and white matter affection, voxel-based morphometry and diffusion tensor imaging are performed, and data are statistically analyzed including (i) group comparisons between patients and controls at baseline and follow-up, and (ii) group comparisons using difference maps to focus on isolated disease-related effects over time.

ELIGIBILITY:
Inclusion criteria for healthy controls:

* written informed consent
* normal neurological examination without any acute or former neurological or severe psychiatric disease, no medical history of traumatic brain injury

Inclusion criteria for patients:

* written informed consent
* diagnosis confirmed by genetic testing
* no other neurological or severe psychiatric disease, no medical history of traumatic brain injury

Exclusion criteria for healthy controls and patients:

* use of psychoactive substances including alcohol (except nicotine), formerly or currently; treatment with modafinil
* severe psychiatric disorders, serious physical illnesses, particularly cardiovascular diseases, formerly or currently
* non-removable ferromagnetic metallic implants, sensors, stimulators, prostheses, pacemaker, large tattoos
* claustrophobia
* age under 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with genetically proven myotonic dystrophy type 1 and myotonic dystrophy type 2 and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2007-05; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in diffusivity indices as assessed by brain MRI with diffusion tensor imaging (DTI) sequences | First analysis at baseline and after 5 years at follow-up
Gray matter changes assessed by magnetic resonance imaging (MRI)-voxel-based morphometry (VBM) | First analysis at baseline and after 5 years at follow-up
Quantification of white matter lesions using age-related white matter changes (ARWMC) rating scale | First analysis at baseline and after 5 years at follow-up

SECONDARY OUTCOMES:
MIRS (Muscular impairment rating scale) | First analysis at baseline and after 5 years at follow-up
  Rating scale to assess disease severity in myotonic dystrophy type 1 patients
Motor performance (Purdue Pegboard, bimanual) | First analysis at baseline and after 5 years at follow-up
  A bimanual task to assess fine motor function in patients and controls. Results are used as a covariate for neuropsychological tests
Beck Depression Inventory (BDI) | First analysis at baseline and after 5 years at follow-up
  To assess depressive symptoms
Boston Naming Test | First analysis at baseline and after 5 years at follow-up
  A test to evaluate semantic memory.
Verbal memory recognition task, a subtest of a computerised neuropsychological screening test battery, named NeuroCogFX (Fliessbach et al., 2006). | First analysis at baseline and after 5 years at follow-up
  Word list learning: 3 repetitions of word list presentation, 12 words. Yes/No recognition test (items:distractors 1 : 2) (reaction intervall: 2 seconds).
  Data measurement: reaction time, number of correct hits
Figural memory recognition task, a subtest of a computerised neuropsychological screening test battery, named NeuroCogFX (Fliessbach et al., 2006). | First analysis at baseline and after 5 years at follow-up
  Figural pattern learning: 12 different checkerboard patterns are presented, 3 repetitions of checkboard pattern presentation. Checkerboard consists of 3x3 fields, each pattern consists of 4 highlighted fields. Yes/No recognition test (items:distractors 1 : 2) (reaction interval: 2 seconds).
  Data measurement: reaction time, number of correct hits
Focussed Attention. Focussed attention concerning processing speed is assessed with a symbol-counting task (subtest 1 of the "Cerebraler Insuffizienztest", c.I.T.S. (Lehrl, 1997)). | First analysis at baseline and after 5 years at follow-up
  Data measurement: time
Psychomotoric Speed. Psychomotoric speed is assessed using the Trail-Making Test, TMT A (Reitan, 1958). | First analysis at baseline and after 5 years at follow-up
  The TMT-A test consists of 25 numbered circles randomly distributed over a sheet of paper. The study participant needs to draw lines to connect the numbers in ascending order.
  Data measurement: time
Reaction time, a subtest of a computerised neuropsychological screening test battery, named NeuroCogFX (Fliessbach et al., 2006). | First analysis at baseline and after 5 years at follow-up
  Data measurement: time
Selective attention (Choice reaction time), a subtest of a computerised neuropsychological screening test battery, named NeuroCogFX (Fliessbach et al., 2006). | First analysis at baseline and after 5 years at follow-up
  Data measurement: time
Interference. Interference is analysed using two tasks. | First analysis at baseline and after 5 years at follow-up
  1. Response inhibition subtest of the "Cerebraler Insuffizienztest" (c.I.T.I; Lehrl and Fischer, 1997).
  2. Inverted choice reaction with reversed conditions of a choice reaction task, a subtest of a computerised neuropsychological screening test battery, named NeuroCogFX (Fliessbach et al., 2006).
  Data measurement: reaction time
Attention shift. Attentional shift is analysed using the the Trail-Making Test, TMT B (Reitan, 1958). | First analysis at baseline and after 5 years at follow-up
  The TMT B test consists of 25 circles randomly distributed over a sheet of paper. These circles include both numbers and letters. The study participant needs to draw lines to connect the numbers and letters in an ascending order, but alternating between numbers and letters.
  Data measurement: time
Visual-spatial / visual-constructive abilities. Visual-spatial / visual-constructive abilities are investigated using the Block design Test (part of "Hamburg-Wechsler Intelligenztest für Erwachsene"-Revision (HAWIE-R); Tewes, 1991). | First analysis at baseline and after 5 years at follow-up
  The block design test consists of 9 blocks and 9 pictures. The study participant needs to look at the picture and reconstruct each picture by arranging all 9 blocks.
  Data measurement: time
Phonematic fluency. Phonemic verbal word fluency is assessed using the oral word-fluency test, subtest 6 of the "Leistungsprüfsystem"; Horn, 1983. | First analysis at baseline and after 5 years at follow-up
  In a given time (one minute) the study participant needs to list as many words that begin with a certain letter.
  Data measurement: number of correct words
Semantic fluency. Semantic word fluency is assessed using a test by Strauss et al.,2006. | First analysis at baseline and after 5 years at follow-up
  A certain category is provided and in a given time (one minute) the study participant needs to list as many items belonging to that category.
  Data measurement: number of correct items
Daytime Sleepiness Scale (DSS) | First analysis at baseline and after 5 years at follow-up
Krupp's Fatigue Severity Scale (KFSS) | First analysis at baseline and after 5 years at follow-up
Epworth Sleepiness Scale (ESS) | First analysis at baseline and after 5 years at follow-up
Pittsburgh Sleep Quality Index (PSQI) | First analysis at baseline and after 5 years at follow-up
Ullanlinna-Narcolepsy Scale (UNS) | First analysis at baseline and after 5 years at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Kornblum, Prof. Dr., Study Chair — Department of Neurology, University Hospital of Bonn, Bonn, Germany; Bernd Weber, Prof. Dr., Study Chair — Life and Brain Center, Department of NeuroCognition-Imaging, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided